CLINICAL TRIAL: NCT01134432
Title: Anti-CD20 Antibody Rituximab in Addition to Prednisolone in Treatment of Warm Antibody Related Autoimmune Hemolytic Anemia. A Randomised Danish Multicenter Trial.
Brief Title: Prednisolone +/- Addition of Anti-CD20 Antibody, Rituximab, in Patients With Immune Hemolytic Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIHA-KA04062-gms
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Anemia, Hemolytic, Autoimmune
Keywords: autoimmune hemolytic anemia; hemolytic anemia; Rituximab; Treatment of autoimmune hemolytic anemia; warm antibody dependant autoimmune hemolytic anemia
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune; Anemia, Hemolytic | interventions — Prednisolone; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prednisolone + Rituximab (Experimental)
  Interventions: Drug: prednisolone + mabthera
- Prednisolone (Active Comparator)
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: prednisolone + mabthera — Prednisolone: 1,5 mg/kg for two weeks with gradually reduced dosis over two months.
  Mabthera: 375 mg/m2 once a week for four weeks
  Other Names: mabthera equals Rituximab
  Arms: Prednisolone + Rituximab
Drug: Prednisolone — Prednisolone: 1,5 mg/kg for two weeks and then gradually reduced dosis over two months
  Arms: Prednisolone

SUMMARY:
The conventional treatment in warm-antibody dependent autoimmune haemolytic anaemia (AIHA) is high-dose glucocorticoid, but in more than half of the patients, haemolytic activity will recur after end of treatment or during the gradual reduction in dose of the drug. As a result, many patients will finally be splenectomized or be treated with long-term glucocorticoids or other immunosuppressive drugs as azathioprine or cyclophosphamide. Recent studies have shown however, that some patients will respond to treatment with the chimeric anti-CD 20 antibody Rituximab and is some cases, the response is permanent. In most of the studies, Rituximab has been used in refractory disease or at least as second line treatment. In this study, patients with AIHA are randomized to receive either high-dose prednisolone with gradual reduction in dose over 2-3 months alone or in combination with Rituximab 375 mg/m2 once a week for 4 weeks. The efficacy of Rituximab will be evaluated by a comparison of the patients in the two treatment arms. The primary treatment goal is a reduction in the number of patients who obtain long-term complete or partial remission. The secondary treatment goal is a reduction in patients who will be splenectomised or receive other immunosuppressive drugs. Finally a comparison of side effects of the treatments will take place.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or over
* Clinical and biochemical signs of haemolytic anaemia
* Positive Coombs test with anti-IgG on its own or with anti-CD3d
* Adequate contraceptive measures (intrauterine device, contraceptive pill or gestagen deposit) for women of childbearing potential

Exclusion Criteria:

* Performance status > 2
* Previous treatment with Rituximab
* Other immune suppressive or anti neoplastic treatment including prednisolone within 3 months
* Auto immune haemolytic anaemia within 6 months
* Other serious disease
* Pregnant women and nursing mothers. Adequate contraceptive measures must be taken for the duration of the study.
* Contraindication for treatment with Rituximab, i.e. patients that develop hypersensitivity/allergy to the contents of the drug or have antibodies against murine proteins.
* Active infection which requires antibiotic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2005-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Number of patients in each group in complete or partial remission | End of treatment and follow-up for 12 months

SECONDARY OUTCOMES:
Side effects | End of treatment plus follow-up for 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Henrik S Birgens, MD, Principal Investigator — Department of Haematology (L121), Copenhagen University Hospital Herlev
Locations (11):
- Denmark (11):
  - Aalborg Hospital, Aalborg
  - Rigshospitalet - Copenhagen University Hospital, Copenhagen
  - Esbjerg Sygehus, Esbjerg
  - Haderslev Sygehus, Haderslev
  - Department of Haematology, Herlev Hospital, Herlev
  - Holstebro Sygehus, Holstebro
  - Naestved Sygehus, Næstved
  - Odense University Hospital, Odense
  - Roskilde Hospital, Roskilde
  - Vejle Hospital, Vejle
  - Viborg Sygehus, Viborg